CLINICAL TRIAL: NCT01754857
Title: Phase II Study of Bendamustine and Rituximab Induction Chemoimmunotherapy Followed by Maintenance Rituximab and Lenalidomide in Previously Untreated Chronic Lymphocytic Leukemia (CLL) and Small Lymphocytic Lymphoma (SLL)
Brief Title: Bendamustine and Rituximab Induction Therapy and Maintenance Rituximab and Lenalidomide in Previously Untreated CLL/SLL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Celgene Corporation (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO11414; 2017-0072 (Other: HS IRB Number); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); NCI-2013-00485 (Registry Identifier: NCI Trial ID); Protocol Version 3/1/2020 (Other: UW Madison)
Record Dates: First submitted 2012-11-09; First posted 2012-12-21 (Estimated); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Lymphoid Leukemia; Small Lymphocytic Lymphoma; Lymphoma, Non-Hodgkin
Keywords: Lymphoid Leukemia; Bendamustine; Rituximab; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphoid; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — Bendamustine Hydrochloride; Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bendamustine, rituximab, lenalidomide (Experimental): INDUCTION: Bendamustine 90mg/m2 IV D1&2 and rituximab IV D1 (up to day 5 of course 1) every 28 days for 6 cycles. Patients with objective response move to maintenance therapy. Patients with objective response after 4 courses are eligible to for maintenance therapy if ongoing induction therapy is associated w/unacceptable toxicity.
  MAINTENANCE: At 6-12 wks post induction therapy, patients receive rituximab IV on day 1 of odd-numbered cycles for 24 cycles; lenalidomide 5mg PO daily on days 1-21 of each cycle (28 day cycles). Dose escalation to 10mg daily on days 1-21 allowed at start of cycle 2 or at start of subsequent cycles in subjects w/acceptable toxicities. Lenalidomide dose escalation only allowed at start of a new cycle up to a max dose of 10 mg/day on days 1- 21. Subjects entering maintenance with CrCl ≥40 & <60mL/min will begin dosing at 5mg every other day on days 1-21. Patients with excessive toxicity from lenalidomide may continue maintenance therapy with rituximab alone.
  Interventions: Drug: Bendamustine; Drug: Rituximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Bendamustine — Given IV
Drug: Rituximab — Given IV
Drug: Lenalidomide — Given PO

SUMMARY:
The investigators propose a treatment strategy where patients are treated with induction chemoimmunotherapy consisting of rituximab + bendamustine for 6 cycles, followed by initiation of maintenance rituximab and lenalidomide among patients achieving an objective response (i.e., at least stable disease with some tumor shrinkage) to induction therapy. The goal of maintenance therapy will be to capitalize on the cytoreduction following induction chemotherapy with a maintenance regimen that has also shown promising activity in CLL, in order to allow for improved PFS in this population.

DETAILED DESCRIPTION:
This is a phase II single arm, open-label, multicenter study evaluating the efficacy and safety of the combination of induction chemoimmunotherapy with bendamustine and rituximab followed by maintenance therapy with rituximab and lenalidomide in subjects with CLL or SLL who have not received any prior cytotoxic chemotherapy for their disease (i.e., prior single-agent rituximab is permitted). The study will be carried out at the University of Wisconsin Carbone Cancer Center (UWCCC).

The subject participation will include a screening period, treatment period, and a follow-up period. The treatment period will extend from the first dose of study drug treatment (day 1, cycle 1 of induction chemoimmunotherapy) until any of the following: completion of the entire course of induction and maintenance therapy; progressive disease (PD); an unacceptable adverse event (AE); the initiation of alternate anti-neoplastic therapy; or a decision by the subject or by the investigator to discontinue treatment; or death. The induction chemoimmunotherapy regimen consists of bendamustine and rituximab for 6 cycles, followed by initiation of maintenance therapy with rituximab and lenalidomide among subjects achieving an objective response to induction therapy (i.e., complete or partial response; stable disease with objective evidence of tumor shrinkage). Subjects with objective response after 4 cycles of bendamustine + rituximab (BR) are eligible to proceed to maintenance therapy if toxicities are limiting further BR induction therapy, or if the treating physician determines that further BR induction therapy would be associated with excessive risk for additional toxicities.

To minimize toxicity with induction chemotherapy, we have chosen a dose of bendamustine at 90 mg/m2/day on days 1 & 2 every 28 days for a total of 6 cycles. Rituximab will be administered at a dose of 500 mg/m2 IV on day 1 of each cycle of induction chemoimmunotherapy (375 mg/m2 cycle 1 only); however, patients at high-risk for cytokine release syndrome may receive rituximab on day 2 of induction therapy. In select circumstances in subjects at high risk for cytokine release syndrome and/or tumor lysis syndrome, rituximab may be administered as late as day 5 of cycle 1 (this alternative dosing of rituximab applies to cycle 1 of induction therapy only). Lenalidomide and rituximab maintenance will be initiated 6-12 weeks after the 6th cycle of chemotherapy, and continued for a total of 24 cycles. Maintenance therapy will continue for a maximum of 24 cycles or until unacceptable toxicity or progression of disease.

Maintenance therapy will begin once there has been adequate hematologic recovery (ANC ≥1000/µL and platelets ≥50,000/µL) and other criteria as outlined in Section 7.5 have been met. Rituximab will be administered at a dose of 375 mg/m2 IV on day 1 of every odd-numbered 28 day cycle (cycles 1,3,5,7,9,11,13,15,17,19,21,23) for a maximum of 12 doses during the maintenance phase. Subjects will receive concurrent lenalidomide 5 mg orally daily on days 1-21 of cycles 1-24 (28 day cycles). If subjects do not experience adverse effects from lenalidomide, dose escalation up to 10 mg orally daily on days 1-21 of each 28 day cycle will be allowed at the start of cycle 2 or at the start of any subsequent cycle (see Section 9.2.3 and 9.2.5 for criteria required to escalate the dose of lenalidomide to 10 mg/day on days 1-21). Lenalidomide dose escalation is only allowed at the start of a new cycle to a maximum dose of 10 mg/day on days 1-21. Subjects entering maintenance with reduced renal function (i.e., creatinine clearance ≥40 but <60 mL/min) will start lenalidomide at a dose of 5 mg every other day. There is no dose modification of rituximab based on reduced renal function. Among subjects without excessive toxicity or evidence of progression, treatment with lenalidomide will continue for up to 24 cycles (cycle 1-24) and treatment with rituximab will continue for up to 12 doses (administered every odd-numbered cycle during cycles 1,3,5,7,9,11,13,15,17,19,21,23). If subjects have excessive toxicity from lenalidomide, ongoing maintenance therapy with rituximab alone is permitted after lenalidomide is discontinued. After completing 24 cycles of maintenance therapy, subjects will then be observed for evidence of PD with clinical assessments every 3 months for at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL)
* No prior cytotoxic chemotherapy for their disease; prior therapy with single-agent rituximab is permitted
* Understand and voluntarily sign an informed consent document
* In cases of SLL, subjects must have at least one bidimensionally measurable lesion at least >= 1.5 cm measured in one dimension
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2 at study entry
* Absolute neutrophil count >= 1500/uL
* Platelet count >= 100,000/uL
* Subjects with neutrophils < 1500/uL or platelets < 100,000/uL with splenomegaly or extensive bone marrow involvement as the etiology for their cytopenias are eligible
* Subjects must have adequate renal function with a creatinine clearance of >= 40 mL/min as determined by the Cockcroft-Gault calculation
* Total bilirubin =< 2 x upper limit laboratory normal (ULN); subjects with non-clinically significant elevations of bilirubin due to Gilbert's disease are not required to meet these criteria
* Serum transaminases aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5 x ULN
* Serum alkaline phosphatase =< 5 x ULN
* Disease-free of prior malignancies for >= 2 years with the exception of basal or squamous cell skin carcinoma, carcinoma "in situ" of the breast or cervix, or localized prostate cancer (treated definitively with hormone therapy, radiotherapy, or surgery)
* Life expectancy of at least 3 months
* All study participants must be willing to be registered into the mandatory Revlimid REMS program after completion of induction chemoimmunotherapy and prior to maintenance therapy, and be willing and able to comply with the requirements of the Revlimid REMS program
* Subjects must not have a known history of hypersensitivity to mannitol
* Prior therapy with rituximab is permitted, even in the setting of rituximab-refractory disease
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS program
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (subjects intolerant to aspirin may use warfarin or low molecular weight heparin) if clinically indicated
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for cycle 1 (prescriptions must be filled within 7 days as required by the Revlimid REMS® program) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent document or complying with the protocol treatment
* Pregnant or breast-feeding females; lactating females must agree not to breast-feed while taking lenalidomide
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Subjects are not eligible if there is a prior history or current evidence of central nervous system or leptomeningeal involvement
* Known hypersensitivity to thalidomide
* Concurrent use of other anti-cancer agents or treatments
* Known to be positive for human immunodeficiency virus (HIV) or infectious hepatitis (type B or C)
* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical or breast cancer, or other cancer from which the subject has been disease free for at least 2 years
* Severe or life-threatening anaphylaxis or hypersensitivity reaction when previously exposed to rituximab or other monoclonal antibody therapy
* Chronic hepatitis B or hepatitis C infection
* New York Heart Association class 3-4 heart failure
* More than one grade 2 or higher transaminase elevation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-11-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Chang, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Chang JE, Havighurst T, Kim K, Eickhoff J, Traynor AM, Kirby-Slimp R, Volk LM, Werndli J, Go RS, Weiss M, Blank J, Kahl BS. Bendamustine + rituximab chemoimmunotherapy and maintenance lenalidomide in relapsed, refractory chronic lymphocytic leukaemia and small lymphocytic lymphoma: A Wisconsin Oncology Network Study. Br J Haematol. 2016 Apr;173(2):283-91. doi: 10.1111/bjh.13957. Epub 2016 Feb 23. PMID 26913697
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Bendamustine, Rituximab, Lenalidomide: INDUCTION: Bendamustine 90mg/m2 IV D1&2 and rituximab IV D1 (up to day 5 of course 1) every 28 days for 6 cycles. Patients with objective response move to maintenance therapy. Patients with objective response after 4 courses are eligible to for maintenance therapy if ongoing induction therapy is associated w/unacceptable toxicity.
  MAINTENANCE: At 6-12 wks post induction therapy, patients receive rituximab IV on day 1 of odd-numbered cycles for 24 cycles; lenalidomide 5mg PO daily on days 1-21 of each cycle (28 day cycles). Dose escalation to 10mg daily on days 1-21 allowed at start of cycle 2 or at start of subsequent cycles in subjects w/acceptable toxicities. Lenalidomide dose escalation only allowed at start of a new cycle up to a max dose of 10 mg/day on days 1- 21. Subjects entering maintenance with CrCl ≥40 & <60mL/min will begin dosing at 5mg every other day on days 1-21. Patients with excessive toxicity from lenalidomide may continue maintenance therapy with rituximab alone.
  Bendamustine: Given IV
  Rituximab: Given IV
  Lenalidomide: Given PO
Period: Overall Study
Arm/Group | Bendamustine, Rituximab, Lenalidomide
Started | 36
Completed | 17
Not Completed | 19
Not completed — Adverse Event | 7
Not completed — Disease progression | 3
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 3
Not completed — other complicating disease | 1
Not completed — ineligible to continue onto maintenance | 1
Not completed — Patient does not wish to be treated, but will continue to be followed for survival | 1
Not completed — Patient decided not to begin maintenance therapy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bendamustine, Rituximab, Lenalidomide
Number analyzed (Participants) | 36
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 1
  50-59 years | 7
  60-69 years | 19
  70-79 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: The primary objective is progression-free survival (PFS). Tumor measurements and disease assessments will be performed at the time of screening, following cycles 3 and 6 of induction chemotherapy, every 4 cycles during the maintenance portion of treatment, and at the end of treatment (EOT). Subjects with clinical evidence of progression prior to a planned disease assessment will be evaluated at the time of clinically suspected progression. Follow-up visits for disease assessment will occur every 3 months after the EOT visit until PD, initiation of alternate anti-neoplastic therapy, decision by the subject to withdraw from the study, or death. The follow-up period will begin after the EOT visit, and all subjects will be followed for at least 2 years after completion of therapy or until death or progression and until the last patient has been followed for at least 1 year following completion of therapy.
Time Frame: At least 24 months following completion of therapy, an average of 5 years
Population: Time to progression, for which only 30 patients were assessable due to being off study prior to study timepoint
Measure: Median (90% Confidence Interval); unit: years
Arm/Group | Bendamustine, Rituximab, Lenalidomide
Number analyzed (Participants) | 30
years | 4.76 [3.95 to 5.57]

2. Secondary Outcome: Objective Response Rates
Description: To determine objective response rates (CR + PR). As described in the primary objective, formal disease assessments including imaging will be performed after cycles 3 and 6 of induction chemotherapy and every 4 cycles during the maintenance portion of treatment. Response and progression in cases of SLL will be evaluated using the International Working Group Criteria30 for response in lymphoma. Response and progression in cases of CLL will be evaluated in this study using the Revised IWCLL Criteria31 for response in CLL. Radiological methodologies, techniques and/or physical examination, established at baseline for the assessment and measurement of each identified lesion will be used for all subsequent assessments.
Time Frame: Up to 30 months
Population: Objective response rate to maintenance, for which only 30 patients were assessable due to being off study prior to study timepoint
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine, Rituximab, Lenalidomide
Number analyzed (Participants) | 30
Participants
  Complete response | 12
  Partial response | 18

3. Secondary Outcome: Count of Events Related to Toxicity
Description: To determine toxicities observed with induction chemotherapy and maintenance therapy. Safety evaluations will be based on the incidence, intensity, and type of adverse events (AEs) and clinical laboratory results. Drug doses will be modified as required based on toxicity as assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 4.0.
Time Frame: Up to 30 months
Measure: Number; unit: toxicity related events
Arm/Group | Bendamustine, Rituximab, Lenalidomide
Number analyzed (Participants) | 36
toxicity related events
  Serious Adverse Events due to toxicities | 41
  Adverse Events due to toxicities | 167

ADVERSE EVENTS:
Time Frame: 30 months
Arm/Group | Bendamustine, Rituximab, Lenalidomide
All-Cause Mortality (participants affected / at risk) | 3/36
Serious Adverse Events (participants affected / at risk) | 36/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine, Rituximab, Lenalidomide (N=36)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (6)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 2 (2)
Bronchial infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
GGT increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 26 (26)
Platelet count decreased (Investigations) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 (18)
Depression (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine, Rituximab, Lenalidomide (N=36)
Nausea (Gastrointestinal disorders) | 26 (51)
Constipation (Gastrointestinal disorders) | 24 (41)
Diarrhea (Gastrointestinal disorders) | 24 (53)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 13 (21)
Abdominal pain (Gastrointestinal disorders) | 6 (7)
Vomiting (Gastrointestinal disorders) | 6 (11)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 32 (59)
General disorders and administration site conditions - Other, specify (General disorders) | 14 (54)
Infusion related reaction (General disorders) | 12 (14)
Edema limbs (General disorders) | 11 (15)
Chills (General disorders) | 5 (7)
Fever (General disorders) | 4 (7)
Non-cardiac chest pain (General disorders) | 4 (4)
Pain (General disorders) | 4 (5)
Localized edema (General disorders) | 3 (5)
Flu like symptoms (General disorders) | 2 (3)
Irritability (General disorders) | 2 (2)
Malaise (General disorders) | 2 (2)
Gait disturbance (General disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 29 (117)
White blood cell decreased (Investigations) | 23 (97)
Lymphocyte count decreased (Investigations) | 21 (111)
Platelet count decreased (Investigations) | 13 (24)
Aspartate aminotransferase increased (Investigations) | 5 (7)
Creatinine increased (Investigations) | 4 (7)
Weight loss (Investigations) | 4 (13)
Alanine aminotransferase increased (Investigations) | 3 (3)
Alkaline phosphatase increased (Investigations) | 3 (5)
Blood bilirubin increased (Investigations) | 3 (4)
Investigations - Other, specify (Investigations) | 3 (3)
Weight gain (Investigations) | 3 (3)
GGT increased (Investigations) | 1 (1)
Haptoglobin decreased (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count increased (Investigations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 16 (31)
Infections and infestations - Other, specify (Infections and infestations) | 10 (16)
Sinusitis (Infections and infestations) | 9 (14)
Skin infection (Infections and infestations) | 8 (9)
Lung infection (Infections and infestations) | 5 (15)
Enterocolitis infectious (Infections and infestations) | 4 (6)
Phlebitis infective (Infections and infestations) | 3 (5)
Urinary tract infection (Infections and infestations) | 3 (4)
Bronchial infection (Infections and infestations) | 2 (3)
Otitis media (Infections and infestations) | 2 (2)
Paronychia (Infections and infestations) | 2 (2)
Penile infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (2)
Tooth infection (Infections and infestations) | 1 (3)
Vaginal infection (Infections and infestations) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 19 (43)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 13 (26)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (13)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 16 (26)
Dizziness (Nervous system disorders) | 11 (15)
Dysgeusia (Nervous system disorders) | 9 (9)
Paresthesia (Nervous system disorders) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4)
Nervous system disorders - Other, specify (Nervous system disorders) | 2 (3)
Tremor (Nervous system disorders) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (23)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 10 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 8 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (21)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (9)
Hypokalemia (Metabolism and nutrition disorders) | 4 (7)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 12 (14)
Agitation (Psychiatric disorders) | 3 (4)
Anxiety (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 3 (6)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Hypertension (Vascular disorders) | 6 (13)
Phlebitis (Vascular disorders) | 6 (9)
Hot flashes (Vascular disorders) | 5 (5)
Hematoma (Vascular disorders) | 3 (3)
Flushing (Vascular disorders) | 2 (3)
Thromboembolic event (Vascular disorders) | 2 (2)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 9 (29)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (7)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (3)
Eye disorders - Other, specify (Eye disorders) | 5 (5)
Conjunctivitis (Eye disorders) | 4 (5)
Dry eye (Eye disorders) | 3 (3)
Blurred vision (Eye disorders) | 2 (3)
Cataract (Eye disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (25)
Urinary frequency (Renal and urinary disorders) | 5 (6)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 3 (5)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 3 (8)
Cytokine release syndrome (Immune system disorders) | 2 (2)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT01754857/Prot_SAP_000.pdf